CLINICAL TRIAL: NCT01853917
Title: Evaluation of Barriers to Postpartum Care in HIV Infected Women
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Tanvir K. Bell, MD, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-11-0503
Record Dates: First submitted 2012-06-19; First posted 2013-05-15 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infection; Pregnancy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionaires and structured interview: HIV infected women who are pregnant and receiving care in Harris County Hospital District single arm study Single arm study
  Interventions: Other: questionaires and structured interviews

INTERVENTIONS:
Other: questionaires and structured interviews — We will do questionaires on pregnant women before they have their baby and after they have their baby. We will do structured interviews after they have their baby

SUMMARY:
The purpose of this study is to evaluate why the majority of HIV infected women in the Harris County Health District system who are pregnant do not come to clinic for their HIV disease after they have a baby through questionaires administered prepartum and questionaires and structured interviews postpartum. The study will ask subjects questions about HIV, drug use, depression and social problems.

DETAILED DESCRIPTION:
This study is evaluating information pre and postpartum to assess what are barriers to patients coming into care for HIV after they have a baby. We will try to evaluate recurrent themes in questionaires and interviews to try and identify the barriers to care.

ELIGIBILITY:
Inclusion Criteria: HIV infected pregnant women who

* HIV-infected women who are pregnant by confirmatory tests or an HIV positive woman who has had a baby within the last 6 months and is coming to care postpartum.
* Women who intend to get care at Harris County Hospital District.
* Subjects must be >18 years old.

Exclusion Criteria:

* Women unable to complete questionnaires.
* Women who are unable to speak, read, or understand English or Spanish.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
evaluate results from qualitative interviews | women seen after they have their baby
  we will ask and record responses and enter into an NIVIVO program to evaluate for emergent themes

SECONDARY OUTCOMES:
evaluate results from questionaires | before they have a baby and after they have a baby
  we will evaluate responses from questionaires There will be 8 areas that there are questionnaires about. These include basic information about yourself, about stress, about your support system, about your sense of control, about tobacco use, about for alcohol/drug use, about taking your HIV medications, and about depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvir Bell, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Harris County Hospital District Clinics-Thomas Street Clinic, Northwest Clinic, Houston, Texas
  - Harris County Hospital District Clinics-LBJ hospital, Houston, Texas